CLINICAL TRIAL: NCT01735240
Title: An Open-label, Fixed-sequence, Single-centre Phase I Study to Assess the Effect of Ketoconazole on the Pharmacokinetics of AZD5069 After Oral Administration of a Single Dose AZD5069 to Healthy Male Volunteers
Brief Title: Phase I Study to Assess the Effect on Healthy Male Volunteers of Ketoconazole on the Pharmacokinetics of a Single Dose of AZD5069 Administered Orally.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D3550C00011
Record Dates: First submitted 2012-11-20; First posted 2012-11-28 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Asthma,; Pharmacokinetics,; Cmax,; Tmax,; λz,; AUC,; Ketoconazole,; Metabolite
Keywords: Phase I,; healthy volunteers,; fixed-sequence,; open-label,; ketoconazole,; combination,; safety
MeSH Terms: conditions — Asthma | interventions — N-(2-(2,3-difluoro-6-benzylthio)-6-(3,4-dihydroxybutan-2-yloxy)pyrimidin-4-yl)azetidine-1-sulfonamide; Ketoconazole

ARMS (1):
- First AZD5069, then Ketoconazole + AZD5069 (Experimental): AZD5069 in first period (on 1 day) and in second period (after wash out) ketoconazole alone (on 2 days) then ketoconazole + AZD5069 (on 1 day), then again ketoconazole alone (on 2 days)
  Interventions: Drug: AZD5069; Drug: Ketoconazole

INTERVENTIONS:
Drug: AZD5069 — AZD5069 15 mg (3x5 mg capsules) single administration
Drug: Ketoconazole — Ketoconazole 400 mg (2x200 mg tablets)

SUMMARY:
The main purpose of the study is to compare the change of the AZD5069 Pharmacokinetic profile when administered with ketoconazole. Subjects will be treated first with AZD5069 only followed by a washout period before starting with the combined treatment (both ketoconazole and AZD5069).

DETAILED DESCRIPTION:
An open-label, fixed-sequence, single-centre phase I study to assess the effect of ketoconazole on the pharmacokinetics of AZD5069 after oral administration of a single dose AZD5069 to healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18 to 50 years (inclusive).
* Veins suitable for cannulation or repeated venipuncture.
* Healthy volunteers with neutrophil counts within the laboratory normal reference range at Screening
* Body mass index (BMI) ≥18.0 and ≤30.0 kg/m2 calculated from height and weight at screening; minimum weight 50 kg and maximum weight 100 kg.
* Non-smokers or ex-smokers with no smoking history for the last 3 months prior to screening and a smoking history of less than 10 pack years (1 pack year = tobacco consumption corresponding to 20 cigarettes smoked per day for 1 year) at screening.

Exclusion Criteria:

* Healthy volunteers with latent tuberculosis as suggested by their history and judged by the Investigator
* Healthy volunteers who belong to a high-risk group for HIV infection.
* Known or suspected history of significant drug abuse as judged by the Investigator.
* History of alcohol abuse or excessive intake of alcohol as judged by the Investigator.
* Plasma donation within 1 month of screening or any blood donation/blood loss >500 mL during the 3 months and/or 1350 mL within the 12 months prior to screening.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of AZD5069 (15 mg) and a metabolite (AZ13587715) measured by AUC, AUC(0-t), Cmax, λz, t½λz, tmax, CL/F (AZD5069 only), Vz/F (alone and in combination with Ketoconazole) | Day 1, Day 2 at 24 hours post dose and Day 3 at 48 hours post dose in period 1 and Day 1, 2, 3 at 48 hours post dose and Day 4 at 72 post dose in period 2.
  (AUC(0-t)) area under the plasma concentration-time curve from time zero to time of last quantifiable concentration, (Cmax) observed maximum plasma concentration, (λz) terminal rate constant, (t½λz) terminal half-life, (tmax) time to reach maximum plasma concentration (tmax), (CL/F) apparent oral clearance (AZD5069 only), (Vz/F) apparent volume of distribution.
Pharmacokinetics of Ketoconazole measured by AUC(0-t) and Cmax (in combination with AZD5069) | Day 1, 2, 3 at 48 hours post dose and Day 4 at 72 post dose in period 2.

SECONDARY OUTCOMES:
Numbers of circulating neutrophil in blood measured by AZD5069 administration alone and in combination with Ketoconazole | Day 1, 2, 3 at predose, 4, 8, 12, 24, 48 hours post dose in period 1 and Day 1, 2, 3, 4 at predose, 4, 8, 12, 24, 48 hours post dose
Safety of AZD5069 (15 mg) in combination with Ketoconazole by assessing a panel of adverse events measures: laboratory assessments, vital signs, physical examination and 12-led electrocardiogram. | Up to 2 months
  Measures: laboratory assessments (clinical chemistry, haematology, urinalysis), vital signs (blood pressure, pulse rate, including body temperature), physical examination and 12-led electrocardiogram.

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Larsson, Dr., Study Director — AstraZeneca Pharmaceutical; Gillian Pilbrow, Study Chair — AstraZeneca Pharmaceutical; Leonard Siew, DR., Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital
Locations (1):
- London, United Kingdom

REFERENCES:
- [Derived] Cullberg M, Arfvidsson C, Larsson B, Malmgren A, Mitchell P, Wahlby Hamren U, Wray H. Pharmacokinetics of the Oral Selective CXCR2 Antagonist AZD5069: A Summary of Eight Phase I Studies in Healthy Volunteers. Drugs R D. 2018 Jun;18(2):149-159. doi: 10.1007/s40268-018-0236-x. PMID 29856004
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1339&filename=D3550C00011_Study_Synopsis.pdf